CLINICAL TRIAL: NCT04987697
Title: A Pilot Study of RISE (Resilience, Insight, Self-Compassion, Empowerment) for Nurse Managers
Brief Title: A Pilot Study of RISE for Nurse Managers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: AdventHealth (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 1504917
Record Dates: First submitted 2020-03-03; First posted 2021-08-03 (Actual); Last update posted 2022-02-28 (Actual); Status verified 2022-02

CONDITIONS: Self Compassion; Stress; Burn-Out
MeSH Terms: conditions — Burnout, Psychological | interventions — Counseling

STUDY DESIGN:
Intervention Model Description: Pilot Study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Counseling and Surveys (Other): nine 90-minute weekly psychoeducational group sessions facilitated by a licensed mental health counselor (LMHC).
  Interventions: Behavioral: counseling

INTERVENTIONS:
Behavioral: counseling — nine 90-minute weekly psychoeducational group sessions facilitated by a licensed mental health counselor (LMHC).

SUMMARY:
The purpose of this study is to determine whether RISE for Nurse Managers has a significant impact on nurse managers' post-traumatic growth, resilience, insight, self-compassion, and empowerment, as well as mental well-being, in their personal lives and their working environment.

ELIGIBILITY:
Inclusion Criteria:

1. Adult ≥ 18 years old
2. Licensed as an RN
3. Nurse manager employed by AdventHealth in a hospital-based setting at the Altamonte Springs, Apopka, Carrollwood, Celebration, Connerton, Dade City, Daytona Beach, DeLand, East Orlando, Fish Memorial, Heart of Florida, Kissimmee, Lake Placid, Lake Wales, New Smyrna Beach, North Pinellas, Ocala, Orlando, Palm Coast, Sebring, Tampa, Waterman, Wauchula, Wesley Chapel, Winter Garden, Winter Park, or Zephyrhills campus
4. Able to speak, read, and understand English fluently
5. Able to provide informed consent
6. Willing and able to comply with all study procedures and requirements for the duration of the study

Exclusion Criteria:

1. Employed as a direct care nurse or in another level of nursing leadership (i.e., assistant nurse manager, director of nursing, executive leader)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2021-04-13 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Posttraumatic Growth Inventory | Change from Baseline to 6 months
  21 item questionnaire with a scale of 0-5, with 0 meaning I did not experience this change as a result of my crisis to 5 meaning I experienced this change to a very great degree as a result of my crisis

SECONDARY OUTCOMES:
Brief Cope | Change from Baseline to 6 months
  28 item questionnaire with a scale of 1-4, with 1 meaning I haven't been doing this at all; and 4 meaning I've been doing this a lot
Brief Index of Affective Job Satisfaction | Change from Baseline to 6 months
  4 item questionnaire with a scale of 1-5, with 1 meaning strongly disagree; and 5 meaning strongly agree
Brief Resilience Scale | Change from Baseline to 6 months
  6 item questionnaire with a scale of 1-5, with 1 meaning strongly disagree; and 5 meaning strongly agree
Psychological Empowerment Instrument | Change from Baseline to 6 months
  12 item questionnaire with a scale of A-G, with A meaning very strongly disagree; and G meaning very strongly agree
Perceived Stress Scale | Change from Baseline to 6 months
  10 item questionnaire with a scale of 0-4, with 0 meaning never; and 4 meaning very often
Maslach Burnout Inventory General Survey | Change from Baseline to 6 months
  16 item questionnaire with a scale of 0-6 with 0 meaning never; and 6 meaning everyday
Self-Compassion Scale - Short Form | Change from Baseline to 6 months
  12 item questionnaire with a scale of 1-5, with 1 meaning almost never; and 5 meaning almost always
Self-Reflection and Insight Scale | Change from Baseline to 6 months
  20 item questionnaire with a scale of 1-6; with 1 meaning strongly disagree; and 6 meaning strongly agree

CONTACTS AND LOCATIONS:
Overall Officials: Amanda T Sawyer, PhD, Principal Investigator — AdventHealth
Locations (1):
- AdventHealth Orlando, Orlando, Florida, United States

REFERENCES:
- [Background] Carver CS. You want to measure coping but your protocol's too long: consider the brief COPE. Int J Behav Med. 1997;4(1):92-100. doi: 10.1207/s15327558ijbm0401_6. PMID 16250744
- [Background] Cohen S, Kamarck T, Mermelstein R. A global measure of perceived stress. J Health Soc Behav. 1983 Dec;24(4):385-96. No abstract available. PMID 6668417
- [Background] Kath LM, Stichler JF, Ehrhart MG. Moderators of the negative outcomes of nurse manager stress. J Nurs Adm. 2012 Apr;42(4):215-21. doi: 10.1097/NNA.0b013e31824ccd25. PMID 22441404
- [Background] Kath LM, Stichler JF, Ehrhart MG, Sievers A. Predictors of nurse manager stress: a dominance analysis of potential work environment stressors. Int J Nurs Stud. 2013 Nov;50(11):1474-80. doi: 10.1016/j.ijnurstu.2013.02.011. Epub 2013 Mar 21. PMID 23522937
- [Background] Labrague LJ, McEnroe-Petitte DM, Leocadio MC, Van Bogaert P, Cummings GG. Stress and ways of coping among nurse managers: An integrative review. J Clin Nurs. 2018 Apr;27(7-8):1346-1359. doi: 10.1111/jocn.14165. Epub 2018 Jan 24. PMID 29148110
- [Background] Lee H, Cummings GG. Factors influencing job satisfaction of front line nurse managers: a systematic review. J Nurs Manag. 2008 Oct;16(7):768-83. doi: 10.1111/j.1365-2834.2008.00879.x. PMID 19017239
- [Background] Grant AM, Franklin J, Langford P. The Self-Reflection and Insight Scale: A new measure of private self-consciousness. Social Behavior and Personality. 2002; 30(8): 821-836.
- [Background] Julious SA. Sample size of 12 per group rule of thumb for a pilot study. Pharmaceutical Statistics. 2005; 4(4): 287-291.
- [Background] Maslach C, Jackson SE, & Leiter MP. (1996). Maslach Burnout Inventory manual (3rd ed.). Palo Alto, CA: Consulting Psychologists Press.
- [Background] Raes F, Pommier E, Neff KD, Van Gucht D. Construction and factorial validation of a short form of the Self-Compassion Scale. Clin Psychol Psychother. 2011 May-Jun;18(3):250-5. doi: 10.1002/cpp.702. Epub 2010 Jun 8. PMID 21584907
- [Background] Shirey MR, McDaniel AM, Ebright PR, Fisher ML, Doebbeling BN. Understanding nurse manager stress and work complexity: factors that make a difference. J Nurs Adm. 2010 Feb;40(2):82-91. doi: 10.1097/NNA.0b013e3181cb9f88. PMID 20124961
- [Background] Smith BW, Dalen J, Wiggins K, Tooley E, Christopher P, Bernard J. The brief resilience scale: assessing the ability to bounce back. Int J Behav Med. 2008;15(3):194-200. doi: 10.1080/10705500802222972. PMID 18696313
- [Background] Spreitzer GM. Psychological empowerment in the workplace: Dimensions, measurement, and validation. Academy of Management Journal. 1995; 38(5):1442-1465.
- [Background] Steege LM, Pinekenstein BJ, Arsenault Knudsen E, Rainbow JG. Exploring nurse leader fatigue: a mixed methods study. J Nurs Manag. 2017 May;25(4):276-286. doi: 10.1111/jonm.12464. Epub 2017 Feb 27. PMID 28244184
- [Background] Thompson ER & Phua FTT. A Brief Index of Affective Job Satisfaction. Group & Organization Management. 2012; 37(3): 275-307.
- [Background] Warshawsky NE, Havens DS. Nurse manager job satisfaction and intent to leave. Nurs Econ. 2014 Jan-Feb;32(1):32-9. PMID 24689156
- [Derived] Sawyer AT, McManus K, Bailey AK. A mixed-methods pilot study of a psychoeducational group programme for nurse managers during the COVID-19 pandemic. J Nurs Manag. 2022 Nov;30(8):4126-4137. doi: 10.1111/jonm.13881. Epub 2022 Nov 13. PMID 36326077